CLINICAL TRIAL: NCT00446745
Title: Study of Interaction Between Adipose and Muscle Tissues in the Control of Muscle Mitochondrial Functions
Brief Title: Abdominal Adiposity and Muscle Mitochondrial Functions
Acronym: Mithycal
Status: Completed | Type: Observational
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Responsible Party: Principal Investigator, Yves Boirie, Prof., Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Other Study IDs: AU628
Record Dates: First submitted 2007-03-09; First posted 2007-03-13 (Estimated); Last update posted 2012-09-19 (Estimated); Status verified 2012-09

CONDITIONS: Mitochondrial Respiratory Chain Deficiencies
Keywords: Nutritional and Metabolic Diseases; Insulin resistance; Energy Metabolisms; Skeletal muscle; Visceral Adipose Tissue
MeSH Terms: conditions — Mitochondrial Diseases; Nutritional and Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Abdominal obesity: 60 males were recruited according to waist circumference, from lean to obese values

SUMMARY:
Numerous studies have demonstrated that excess perivisceral adipose tissue is associated with metabolic diseases such as insulin resistance.

In skeletal muscle, insulin resistance has been correlated with reduced mitochondrial oxidative functions. According to the actual theory, mitochondrial dysfunctions are proposed to play a causal role in the aetiology of insulin resistance. Mechanisms involve increased intramyocellular lipids storage. Yet, the causes responsible for the decline in muscle mitochondrial functions remain to be elucidated.

The investigators hypothesize that these alterations are induced by combined changes in plasma profiles of lipids and adipokines, which originate from perivisceral adipose tissue. The study aims at answering the following questions :

* Are muscle mitochondrial functions altered in association with increased perivisceral adipose tissue storage?
* Do changes in the pattern of plasma lipids and adipokines explain this correlation?

DETAILED DESCRIPTION:
Sixty 35 to 50-years old sedentary men will be included based on their abdominal circumference (from 75 to over 102 cm).

Body composition will be evaluated using dual-energy X-ray absorptiometry and perivisceral, intramuscular and intrahepatic adiposity will be assess by MRI and proton-NMR spectroscopy. Subjects will be also characterized by their glucose tolerance (OGTT), basal metabolism (indirect calorimetry) and maximal oxygen consumption (maximal aerobic power test on exercise bike).

Blood samples will be collected in the fasted state to assess lipids and adipokines concentrations.

Biopsies will be obtained from the vastus lateralis muscle to examine mitochondrial functions (respiration rates, ATP and superoxide anion production rates, maximal activity of oxidative enzyme). Gene expression of key enzymes, protein and transcription factors involved in lipid and energy metabolism will be assessed using real-time quantitative PCR.

Finally, whole body and muscle protein metabolism will be investigated in half of the subjects using tracer infusion (incorporation of L-[1-13C]leucine) and biopsies from vastus lateralis, both in the post-absorptive and post-prandial states (test meal)

ELIGIBILITY:
Inclusion Criteria:

* Male subjects
* Age between 35 and 50
* waist circumference > 75 cm
* Baecke score < 1 (activity score for sedentary subjects)
* Subjects giving written informed consent
* Subjects willing to comply with the study procedures
* Subjects considered as normal after clinical examination and medical questionnaire

Exclusion Criteria:

* Weight change > 3 kg within 3 months prior to study
* Patients with type 1 or type 2 diabetes
* Serologic evidence of active hepatitis B or HIV
* History of cancer or significant intestinal, hepatic, renal or cardiovascular disorders within the past 5 years
* History of systemic infections or inflammatory diseases within the past 2 months
* Hypocaloric or special diets (e.g. vegetarian)
* Patients currently known to abuse or to be dependent on any drug, including alcohol (daily consumption > 20g) and tobacco (daily consumption > 5 cigarettes)
* CRP < 5 mg/L
* Blood coagulation disorders
* Allergy to xylocaïne
* for test meal : Food allergy (particularly milk allergy and lactose intolerance)
* for MRI : Claustrophobia

Ages: 35 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * 60 Male subjects
  * Age between 35 and 50
  * waist circumference (Waist) > 75 cm
    15 men with Waist between 75 and <87cm, 15 men with Waist between 87 and <94cm, 15 men with Waist between 94 and <102cm, and 15 men with Waith equal or higher than 102cm.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2006-04; Primary Completion 2006-12 (Actual); Study Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yves Boirie, PU-PH, Principal Investigator — UMR1019 INRA - Auvergne University; Beatrice Morio, PhD, Study Director — UMR 1019 INRA - Auvergne University
Locations (1):
- Centre ed Recherche en Nutrition Humaine d'Auvergne (CRNH), Unité d'Exploration Nutritionnelle, Laboratoire de Nutrition humaine, Clermont-Ferrand, France

REFERENCES:
- [Background] Chanseaume E, Tardy AL, Salles J, Giraudet C, Rousset P, Tissandier A, Boirie Y, Morio B. Chronological approach of diet-induced alterations in muscle mitochondrial functions in rats. Obesity (Silver Spring). 2007 Jan;15(1):50-9. doi: 10.1038/oby.2007.511. PMID 17228031
- [Background] Chanseaume E, Malpuech-Brugere C, Patrac V, Bielicki G, Rousset P, Couturier K, Salles J, Renou JP, Boirie Y, Morio B. Diets high in sugar, fat, and energy induce muscle type-specific adaptations in mitochondrial functions in rats. J Nutr. 2006 Aug;136(8):2194-200. doi: 10.1093/jn/136.8.2194. PMID 16857840
- [Derived] Chanseaume E, Barquissau V, Salles J, Aucouturier J, Patrac V, Giraudet C, Gryson C, Duche P, Boirie Y, Chardigny JM, Morio B. Muscle mitochondrial oxidative phosphorylation activity, but not content, is altered with abdominal obesity in sedentary men: synergism with changes in insulin sensitivity. J Clin Endocrinol Metab. 2010 Jun;95(6):2948-56. doi: 10.1210/jc.2009-1938. Epub 2010 Apr 9. PMID 20382691